CLINICAL TRIAL: NCT04488029
Title: A Parallel, Virtual, Randomized Trial of PCT for Speech, Language, and Cognitive Intervention in Stroke Patients
Brief Title: PCT for Speech, Language, and Cognitive Intervention in Stroke Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Learning Corp (Industry)
Responsible Party: Principal Investigator, Michelle Braley, Primary Investigator/Senior Manager of Clinical Science, The Learning Corp
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLC-PCT-Pilot
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Aphasia, Acquired
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Intervention Model Description: Final study eligibility will be assessed after administration of the Western Aphasia Battery, Revised (WAB-R). Eligible subjects will be pseudorandomly assigned to the experimental group OR the control group, while trying to balance for aphasia severity (WAB-R Aphasia Quotient, WAB-AQ). Subjects in the experimental group will receive therapy via the PCT app during the treatment period. Subjects in the control arm will receive conventional workbook therapy. Subjects in both groups will be asked to refrain from obtaining one-on-one individual aphasia or cognitive therapy. Subjects may participate in organized social groups, such as community aphasia groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): At the start of the study, subjects will be provided with a tablet with videoconferencing software and the PCT app pre-installed. Research staff will remotely setup a PCT account for the subjects, and provide instructions for logging into the PCT application. During the treatment period, patients will be instructed to use PCT for at least 30 minutes a day and at least 5 days a week. Performance data (accuracy and latency) will be reported by the PCT software to the treating clinician and will be used to modify task assignment over time. PCT tracks usage of the program so that research staff can access automated reporting of subject use to monitor participant adherence to the treatment program.
  Interventions: Other: PCT
- Control Group 1 [Conventional Workbook Therapy] (Active Comparator): At the start of the study, subjects will be provided with a tablet with videoconferencing software and the PCT app pre-installed. Subjects in the control group will be told they will have access to 3-months of PCT after their participation in the study has concluded. Subjects in this group will be provided with a standard regime of paper workbooks and instructions to complete approximately 30 minutes a day at least 5 days a week.
  Interventions: Other: Workbooks

INTERVENTIONS:
Other: PCT — PCT is designed to deliver similar therapy as is conventionally provided in-clinic by a Speech Language Pathologist (SLP), which the patient can access from any location using the application installed on a supported tablet. The device functions by allowing clinicians to create a personalized therapy program for each patient from 75 categories of clinical therapies, which patients may access from their tablet device remotely. The PCT software is comprised primarily of authentication and an algorithm that suggests advancement of the therapy program based on observed patient deficits and progress.
  Arms: Experimental Group
Other: Workbooks — Subjects in this group will be provided with a standard regime of paper workbooks (e.g. Workbook for Aphasia: Exercises for Expressive and Receptive Language Functioning; Brubaker, 2006) that are typically used by clinicians to practice therapy tasks with individuals. Notably, the control procedure employed here is similar to that employed on a large-scale study examining technology as a treatment option and involved usual care control group by Palmer and colleagues (2015).
  Arms: Control Group 1 [Conventional Workbook Therapy]

SUMMARY:
Given the evolving uses of technology in rehabilitation, the investigators aimed to measure the change in aphasia severity using PCT App, a digital therapeutic adapted from Constant Therapy (CT), a dynamic, personalized therapy program for people with cognitive, speech, or language disorders.

The entire study, including recruitment, enrollment, assessment and treatment were conducted remotely.

The proposed pilot study seeks to compare performance of PCT therapy vs. conventional workbook intervention for stroke patients. The investigators hypothesize that the experimental (PCT) group will experience greater gains on the WAB-AQ at follow-up compared to baseline compared to a control (workbook) group.

Subjects were prospectively assigned to an experimental or active control group in a random order with both groups balanced for their baseline level of speech, language and/or cognitive ability:

1. Experimental Group: Participants were instructed to use PCT for at least 30 minutes/day, 5 days/week. Performance and usage data were automatically reported by the PCT software to the treating clinician and was used to modify task assignment over time and monitor participant adherence to the treatment program.
2. Active Control Group: Participants were provided with a standard regime of paper workbooks (e.g. Workbook for Aphasia; Brubaker, 2006) that are typically used by clinicians with persons with aphasia (PWA) for at least 30 minutes/day, 5 days/week. Notably, the control procedure employed here is similar to a large-scale study examining technology as a treatment option by Palmer and colleagues (2015).

The treatment period was 10 weeks. All participants received a bimonthly check-in through video-chat with a member of the research staff during the treatment period.

ELIGIBILITY:
Inclusion criteria:

* Have diagnosis of stroke involving a hemorrhage or ischemic event, resulting in speech, language, and/or cognitive deficits
* Have time post-stroke of at least 4 months prior to enrollment
* Have been discharged from rehabilitation hospital
* Are adults (aged 18 years or older) at the time of consent
* Exhibit clinically confirmed speech, language, and/or cognitive deficits based on medical records
* Are fluent English speakers
* Have confirmed aphasia using the WAB-R Aphasia Quotient (score of 90 or lower; 93.8 is cutoff for normal scores)
* Have a presence of a family member or caregiver who is willing and able to provide assistance during the duration of study period

Exclusion Criteria:

* Have comorbid neurological conditions that could impair study participation in the opinion of the investigator, such as dementia or Parkinson's disease
* Currently require inpatient care or acute care
* Are currently undergoing related one-on-one individual therapy at a hospital, rehabilitation facility, university, or at home
* Exhibit severe apraxia of speech or severe dysarthria of speech, as verified by a clinician and confirmed by the WAB-R (and the Screen for Dysarthria and Apraxia of Speech if necessary), and/or medical records
* Have comorbid psychiatric conditions that could impair study participation in the opinion of the investigator, including such as schizophrenia or major depressive disorder, as indicated by medical records
* Have uncorrected hearing or vision loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Western Aphasia Battery Revised, Aphasia Quotient (WAB-AQ) | Baseline assessment
  The WAB-R is a standardized tool that assesses language and cognitive skills and provides scores quantifying the impact of a stroke on those skills. The Aphasia Quotient from the WAB-R includes segments from Part 1 of the assessment, evaluating spontaneous speech including fluency and information content, auditory comprehension, naming, and repetition.
Western Aphasia Battery Revised, Aphasia Quotient (WAB-AQ) | Follow-up assessment 10-12 weeks post baseline
  The WAB-R is a standardized tool that assesses language and cognitive skills and provides scores quantifying the impact of a stroke on those skills. The Aphasia Quotient from the WAB-R includes segments from Part 1 of the assessment, evaluating spontaneous speech including fluency and information content, auditory comprehension, naming, and repetition.

SECONDARY OUTCOMES:
Western Aphasia Battery Revised, Cortical Quotient (WAB-CQ) | Baseline assessment
  The Cortical Quotient as obtained from the WAB-R Parts 1 and 2 was utilized as secondary outcome measures. Part 2 of the WAB-R includes reading, writing, apraxia, constructional, visuospatial, and calculation sections.
Western Aphasia Battery Revised, Cortical Quotient (WAB-CQ) | Follow-up assessment 10-12 weeks post baseline
  The Cortical Quotient as obtained from the WAB-R Parts 1 and 2 was utilized as secondary outcome measures. Part 2 of the WAB-R includes reading, writing, apraxia, constructional, visuospatial, and calculation sections.
Western Aphasia Battery Revised, Language Quotient (WAB-LQ) | Baseline assessment
  The Language Quotient as obtained from the WAB-R Parts 1 and 2 was utilized as secondary outcome measures. Part 2 of the WAB-R informing the Language Quotients includes reading and writing sections.
Western Aphasia Battery Revised, Language Quotient (WAB-LQ) | Follow-up assessment 10-12 weeks post baseline
  The Language Quotient as obtained from the WAB-R Parts 1 and 2 was utilized as secondary outcome measures. Part 2 of the WAB-R informing the Language Quotients includes reading and writing sections.
Brief Test of Adult Cognition by Telephone (BTACT) | Baseline assessment
  The BTACT is a brief, remote, cognitive assessment that evaluates memory for and judgments about words and numbers. It includes tasks such as recall tasks, both immediate and short term, category fluency, and number reasoning and manipulation tasks.
Brief Test of Adult Cognition by Telephone (BTACT) | Follow-up assessment 10-12 weeks post baseline
  The BTACT is a brief, remote, cognitive assessment that evaluates memory for and judgments about words and numbers. It includes tasks such as recall tasks, both immediate and short term, category fluency, and number reasoning and manipulation tasks.
Stroke and Aphasia Quality of Life Scale 39 (SAQOL-39) | Baseline assessment
  The SAQOL-39 is a structured quality of life questionnaire administered to either a patient or a caregiver. It assesses the impact of a stroke on daily activities, communication, emotions, and family and social life by asking patients or caregivers to complete a 5 point rating scale in response to specific questions focusing on the past week alone.
Stroke and Aphasia Quality of Life Scale 39 (SAQOL-39) | Follow-up assessment 10-12 weeks post baseline
  The SAQOL-39 is a structured quality of life questionnaire administered to either a patient or a caregiver. It assesses the impact of a stroke on daily activities, communication, emotions, and family and social life by asking patients or caregivers to complete a 5 point rating scale in response to specific questions focusing on the past week alone.

CONTACTS AND LOCATIONS:
Overall Officials: Swathi Kiran, PhD, CCC-SLP, Study Director — The Learning Corp
Locations (1):
- The Learning Corp, Newton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
De-identified, aggregate only. Data will be available at the request of other investigators for purposes of replicating procedures and results. Anonymized data will be shared by request from any qualified investigator.

REFERENCES:
- [Background] Palmer R, Witts H, Chater T. What speech and language therapy do community dwelling stroke survivors with aphasia receive in the UK? PLoS One. 2018 Jul 10;13(7):e0200096. doi: 10.1371/journal.pone.0200096. eCollection 2018. PMID 29990345
- [Background] Tun PA, Lachman ME. Telephone assessment of cognitive function in adulthood: the Brief Test of Adult Cognition by Telephone. Age Ageing. 2006 Nov;35(6):629-32. doi: 10.1093/ageing/afl095. Epub 2006 Aug 30. No abstract available. PMID 16943264
- [Background] Dekhtyar M, Braun EJ, Billot A, Foo L, Kiran S. Videoconference Administration of the Western Aphasia Battery-Revised: Feasibility and Validity. Am J Speech Lang Pathol. 2020 May 8;29(2):673-687. doi: 10.1044/2019_AJSLP-19-00023. Epub 2020 Mar 19. PMID 32191122
- [Background] Caute A, Northcott S, Clarkson L, Pring T, Hilari K. Does mode of administration affect health-related quality-of-life outcomes after stroke? Int J Speech Lang Pathol. 2012 Aug;14(4):329-37. doi: 10.3109/17549507.2012.663789. Epub 2012 Apr 4. PMID 22472032
- [Derived] Braley M, Pierce JS, Saxena S, De Oliveira E, Taraboanta L, Anantha V, Lakhan SE, Kiran S. A Virtual, Randomized, Control Trial of a Digital Therapeutic for Speech, Language, and Cognitive Intervention in Post-stroke Persons With Aphasia. Front Neurol. 2021 Feb 12;12:626780. doi: 10.3389/fneur.2021.626780. eCollection 2021. PMID 33643204